CLINICAL TRIAL: NCT04181814
Title: Bedside Gastric Ultrasound for Preoperative Assessment of Gastric Content in Diabetic Patients Following ASA Fasting Guidelines
Brief Title: Gastric Ultrasound for Preoperative Assessment of Gastric Content in Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-319
Record Dates: First submitted 2019-11-27; First posted 2019-11-29 (Actual); Last update posted 2020-03-06 (Actual); Status verified 2019-11

CONDITIONS: Aspiration Pneumonia; Gastric Volume
MeSH Terms: conditions — Pneumonia, Aspiration | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Diabetic patients: Diagnosed as diabetes
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Use ultrasound to assess gastric contents in diabetic patients before anesthesia

SUMMARY:
ASA fasting guidelines are only applicable to healthy elective surgery patients. Measuring gastric volume now is not easy, and scintigraphy has remained the gold standard technique for many years. This prospective observational study aim to explore the gastric emptying of type 2 diabetic patients.

DETAILED DESCRIPTION:
ASA fasting guidelines are only applicable to healthy elective surgery patients. Measuring gastric volume now is not easy, and scintigraphy has remained the gold standard technique for many years. Ultrasound has progressively emerged as a useful substitute due to its reduced cost and ease of performance.

Using gastric ultrasound measure gastric antrum cross-sectional area to determine whether patients are empty stomach, help anesthesiologists in preoperative evaluation of diabetic patients with the risk of aspiration, so as to guide the anesthesiologist take effective interventions, this prospective observational study aim to explore the gastric emptying of type 2 diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

1. Ages >18 years old
2. Diabetes (I or II)
3. Following American Society of Anesthesiologists (ASA) fasting guidelines before surgery
4. Undergoing general anesthesia

Exclusion Criteria:

1. Pregnant
2. Gastric Intestinal Tract (GIT) diseases or surgeries affect gastric emptying
3. Diagnosed with liver dysfunction or renal insufficiency
4. Patients who are unable to cooperate or understand the process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic patients undergoing elective surgery and firmly following ASA fasting guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-01-20 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
Gastric contents | before anesthesia
  using ultrasound to evaluate antral cross-sectional area
Risk factors | before anesthesia
  by analysisng full stomach of patients to find risk factors

SECONDARY OUTCOMES:
Perlas grading scale | before anesthesia
  This is a 3-point grading system (grades 0, 1, and 2) based exclusively on qualitative sonographic assessment of the gastric antrum.If a patient's antrum appears empty in both supine and right lateral positions (grade 0), it is likely truly empty. If it appears only mildly distended in the right lateral decubitus position, but not in the supine position (grade 1), the patient likely has a very small volume of gastric fluid within the limits of what is known to be "safe". An antrum that is distended in both supine and right lateral decubitus positions (grade 2) denotes a gastric fluid volume beyond the limits of what is considered safe.

CONTACTS AND LOCATIONS:
Overall Officials: Min Yan, Doctor, Study Chair — The Second Affiliated Hospital of Zhejiang University Medical College
Locations (1):
- The Second Affiliated Hospital of Zhejiang University Medical College, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No